CLINICAL TRIAL: NCT06264141
Title: Multicenter, Randomized, Double-blinded, Placebo-controlled, Phase 2 Clinical Efficacy Study Evaluating Nitric Oxide Nasal Spray (NONS) Compared to Saline Nasal Spray as an Early Treatment for Recurrent Acute Rhinosinusitis (RARS)
Brief Title: Evaluation of Nitric Oxide Nasal Spray (NONS) for Treatment of Recurrent Acute Rhinosinusitis
Acronym: NONS-RARS-01
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sanotize Research and Development corp. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NONS-RARS-01
Record Dates: First submitted 2024-01-23; First posted 2024-02-16 (Actual); Last update posted 2025-01-06 (Actual); Status verified 2024-08

CONDITIONS: Recurrent Acute Rhinosinusitis
Keywords: Sinusitis; Nitric oxide; RARS; NONS; Nasal spray; Rhinosinusitis; Recurrent; Acute
MeSH Terms: conditions — Sinusitis; Rhinosinusitis; Recurrence

STUDY DESIGN:
Intervention Model Description: A two-week therapy of NONS vs Placebo (saline nasal spray) initiated immediately after the onset of a new RARS episode to assess the acceleration to clinical success (cured/much-improved symptoms), lack of use of INCS (Day 5, or thereafter) and rescue oral antibiotics (ATBs) (Day 8, or thereafter) after initiation of nitric oxide-releasing solution (NORS) platform therapy.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: A blinded participant number will be assigned to each randomized participant. Site staff/ physician will then dispense a kit labelled with the authorization number generated during randomization to the individual participant. No study investigators, associates performing assessments or participants will be aware of the study medication in the assigned treatments.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nitric Oxide Releasing Solution (Active Comparator): Nasal spray with nitric oxide releasing solution (NORS) delivered five times per day spaced 1 to 4 hours between each dose while awake.
  Maximum volume delivered: 0.56 mL NORS @ 0.11ppm*hrs
  Interventions: Drug: Nitric Oxide Releasing Solution
- Placebo (Placebo Comparator): Nasal spray with isotonic saline delivered five times per day spaced 1 to 4 hours between each dose while awake.
  Maximum volume delivered: 0.56 mL Saline @ 0.9%
  Interventions: Device: Nasal spray with isotonic saline

INTERVENTIONS:
Drug: Nitric Oxide Releasing Solution — The Sponsor designed a dual chamber nasal spray bottle for NORS administration. Components are mixed from two chambers to create the final NO-producing formulation. The liquid contains NO at 0.11 ppm*hour, which acts as a viricidal agent. Instructions for storing, preparing, and administering the study treatment will be provided to participants.
  Other Names: Nitric Oxide Nasal Spray
  Arms: Nitric Oxide Releasing Solution
Device: Nasal spray with isotonic saline — The Sponsor designed a dual-chamber nasal spray bottle for NORS administration. The bottle will be filled with normal saline before being provided to the participant.
  Other Names: Normal saline, 0.9% saline
  Arms: Placebo

SUMMARY:
A two-week therapy of nitric oxide nasal spray (NONS) vs Placebo (saline nasal spray) initiated immediately after the onset of a new Recurrent Acute Rhinosinusitis (RARS) episode to assess the acceleration to clinical success (cured/much improved symptoms), lack of use of intranasal corticosteroids (INCS) (Day 5, or thereafter) and rescue oral antibiotics (ATBs) (Day 8, or thereafter) after initiation of nitric oxide releasing solution (NORS) platform therapy.

DETAILED DESCRIPTION:
Study Design:

This is a multicenter, randomized, double-blind placebo-controlled, two-arm, parallel-group, phase 2 clinical trial to determine the efficacy and safety of NONS to treat recurrent acute (bacterial) rhinosinusitis (RARS).

Nitric oxide-releasing solution (NORS) therapy administered as NONS, has the potential to shorten RARS episodes and may reduce the concomitant use of INCS, oral non-steroidal anti-inflammatory drugs (NSAIDS) and oral ATBs used to manage this condition. Suitable candidates will be randomized to a 2-week course of nitric oxide nasal spray (NONS) compared to saline nasal spray (1:1 ratio, administered as five doses daily). RARS symptoms efficacy response will be measured twice daily, after initiation of study medication (Day 1 to Day 15), then once daily to the end of the study (Day 16 to Day 29). The goal of NONS therapy is to accelerate the time to achieve RARS symptoms resolution, defined as a clinical success (cured or much improved sinusitis symptoms; primary endpoint assessment at Day 8), minimize the use of INCS and the avoidance of rescue oral ATBs (both secondary endpoints) over the study period (Day 1 to Day 29). Participants will be enrolled between RARS episodes while asymptomatic, and on study for up to 4 months or until their next recurrence of RARS at which time study procedures and medication begin.

Adults (18 years or older) presenting with a history of mild to severe RARS symptoms (nasal obstruction (congestion), purulent nasal discharge, postnasal drip, headache, facial pain), signs (such as facial swelling), and other nonspecific signs/symptoms of fever and malaise are eligible.

The primary endpoint is is the time to sinus symptoms resolution, i.e., being cured or much improved (participant reported clinical success) after 7 days of therapy,

ELIGIBILITY:
Inclusion Criteria:

1. At least aged 18 years old at the time of consent (19 years depending on the age of majority in the Canadian province/territory).
2. History of recurrent acute bacterial sinusitis (ABS) with at least three episodes in the previous 12 months with at least two episodes requiring ATB therapy (with symptom-free periods between infections).
3. History of at least two moderately severe symptoms of acute rhinosinusitis (anterior (nasal) and posterior (postnasal drip) secretions, nasal obstruction (congestion), headache or facial pain/pressure during a typical RARS episode.
4. If female, be surgically sterile or post-menopausal (no menses for at least 12 months), or if of childbearing potential, must be using an acceptable method of contraception such as a combination estrogen/progestin hormonal contraceptive (oral or injected) for at least 1 month prior to Screening, or such items as an intrauterine device (IUD), intrauterine system (IUS), transdermal hormonal implant, vaginal hormonal ring, or 2 forms of the following: diaphragm, cervical cap, patch, condom, spermicide, or sponge. Total abstinence is permitted. Must agree to agree continue using contraception for the duration of the study medication treatment.
5. If male, be surgically sterile, or agree to use appropriate contraception (latex condom with spermicide) when engaging in sexual activity and agree to not donate sperm for the duration of the study medication treatment.
6. Be reasonable stable health (i.e., diagnosed chronic illnesses that are not deemed stable by the participant's primary care physician), or in the opinion of the Investigator, based on medical history (i.e., absence of any clinically relevant abnormality) during Screening.
7. Be able to understand and provide written, informed consent.
8. Must be able to attend on-site and virtual study visits.

Exclusion Criteria:

1. Complicated RARS (orbital or intracranial involvement).
2. Symptoms attributed to sinus disease for longer than 4 weeks.
3. RARS with multiple courses of antimicrobial therapy failures (in previous 2 years, 3 or more episodes treated with 2 or more ATBs).
4. Disease history consistent with severe allergic or seasonal rhinitis (requiring oral cortico-steroids to manage intractable nasal symptoms).
5. Isolated frontal and sphenoidal clinical disease (given the different pathophysiology and etiologic pathogens).
6. History of nasal polyposis.
7. History of abnormal sinus pathology.
8. Previous sinus surgery.
9. Participants with cystic fibrosis.
10. Recurrent moderate epistaxis.
11. Participants with chronic obstructive pulmonary disease (COPD).
12. Participants with severe asthma (per European Respiratory Society (ERS)/American Thoracic Society (ATS) 2014).
13. Immunocompromised participants or participants with other medical conditions that may affect interpretation of the effect of trial drugs.
14. Allergic to any of the trial drugs.
15. Females who are breastfeeding, pregnant, or attempting to become pregnant.
16. Participants who have conditions that participation is not in their best interest.
17. Participants whose participation in the study, in the opinion of the Investigator, have a condition which would interfere with their ability to adhere to the protocol (e.g., participants whom are mentally or neurologically disabled and whom are considered not fit to their participation in the study), interfere with the assessment of the investigational product, or compromise the safety of the participant or the quality of the data.
18. Participants who are unable to sign the informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 162 (Actual)
Dates: Start 2024-01-16 (Actual); Primary Completion 2025-02-24 (Estimated); Study Completion 2025-02-24 (Estimated)

PRIMARY OUTCOMES:
Primary endpoint is the time to sinus symptoms resolution | 8 days
  To demonstrate superior efficacy of NONS compared to saline nasal spray in the early treatment of RARS. The primary objective is to demonstrate that NONS accelerates the time to achieve clinical success as determined by a higher percentage of participants having resolved or much improved sinusitis symptoms after 7 days of therapy.

SECONDARY OUTCOMES:
Time (days) to full recovery from sinusitis (participant reported) | 29 days
  To record the rate of recovery for study participants.
Time (days) to sinus symptoms resolution, i.e., being cured or much improved (participant reported clinical success) | 29 days
  To record the improvement of symptoms among study participants.
Time (days) to the initiation of rescue oral ATB(s), i.e., treatment failure i.e., treatment failure | 29 days
  To record the frequency of study participants receiving rescue antibiotics.
Time (days) to initiation of INCS | 29 days
  To record the rate of study participants starting corticosteroids.
Proportion of participants requiring INCS | Day 5, 8, 15 & 29
  To record the fraction of study participants requiring corticosteroids.
Proportion of participants requiring rescue oral ATBs | Day 5, 8, 15 & 29
  To record the fraction of study participants requiring antibiotics.
Proportion of participants recovered from sinusitis | Day 5, 8, 15 & 29
  To record the fraction of study participants who recover
Proportion of participants with rapidly worsening symptoms requiring the use of INCS and oral ATBs | 29 days
  To record the fraction of study participants whose symptoms required corticosteroids and antibiotics.
Proportion of participants achieving at least a 9-point improvement change from baseline in Sinonasal Outcome Test (SNOT)-22 | Day 8 & 15
  To record the fraction of study participants who show improvement in survey scores.
Tolerability and safety of NONS | 29 days
  Number of participants with clinically significant changes from baseline in Adverse events
Proportion of participants with clinically significant changes from baseline in vital signs | 29 days
  Vital sign measurements includes systolic/diastolic blood pressures, pulse rate, respiratory rate and body temperature
Proportion of participants with clinically significant changes from baseline in laboratory parameters | 29 days
  Laboratory investigation includes hematology and chemistry panels
Number of participants with clinically significant changes from Baseline in physical examinations | 29 days

OTHER OUTCOMES:
Number of ATB courses required as a rescue treatment | 29 days
  To record the number of antibiotic courses taken by individual participants.
Time (days) to the initiation of NSAIDs | 29 days
  To record the duration to study participants receiving NSAIDs.
Proportion of participants requiring NSAIDs | 29 days
  To record the fraction of participants requiring NSAIDs.
Time (days) to each symptom being cured or much improved | 29 days
  To record the duration to symptom cure/improvement by symptom.
Proportion of participants being cured or much improved for each symptom | Day 8, 15 & 29
  To record the fraction of participants with symptom improvement per each symptom.
Proportion of participants achieving at least a 50% reduction in sinusitis symptoms (by MRSS) | Day 5, 8, 15 & 29
  To record the fraction of participants reporting significant improvement on their major rhinosinusitis symptom score.
  MRSS minimum score value is 0 (no symptoms), maximum score value is 15 (worst symptoms).

CONTACTS AND LOCATIONS:
Overall Officials: Keith Moore, PharmD, Study Director — Sanotize Research and Development corp.
Locations (7):
- Canada (7):
  - Okanegan Clinical Trials, Kelowna, British Columbia
  - Richmond Clinical Trials (Okanagan Clinical Trials Satelite Site), Richmond, British Columbia
  - Cliantha Research, Mississauga, Ontario
  - Clinical Research of Ontario, Scarborough Village, Ontario
  - Intermed Groupe Santé, Chicoutimi, Quebec
  - Alpha Recherche Clinique LeBourneuf, Québec, Quebec
  - Alpha Recherche Clinique Val-Belair, Québec, Quebec